CLINICAL TRIAL: NCT07184931
Title: A Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled Phase 3, Induction Study to Evaluate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: An Induction Study to Investigate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Crohn's Disease
Acronym: STARSCAPE-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18326; 2025-521036-11 (Registry Identifier: CTIS); U1111-1314-5319 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Duvakitug Dose 1 (Experimental): Subcutaneous (SC) Injection as per protocol
  Interventions: Drug: Duvakitug
- Duvakitug Dose 2 (Experimental): SC injection as per protocol
  Interventions: Drug: Duvakitug
- Placebo (Placebo Comparator): SC injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duvakitug — Pharmaceutical form:Injection solution Route of administration:SC injection
  Other Names: SAR447189
  Arms: Duvakitug Dose 1; Duvakitug Dose 2
Drug: Placebo — Pharmaceutical form:Injection solution Route of administration:SC injection
  Arms: Placebo

SUMMARY:
This is a multinational, multicenter, randomized, double-blind, placebo-controlled, Phase 3 induction study, comprised of 3 sub-studies, to evaluate the efficacy and safety of duvakitug in participants with moderately to severely active CD. Study details include:

The study duration may be up to 35 weeks with:

* Up to 5-week Screening Period.
* 12-week Sub-Study 1 (Single Arm Open-Label Feeder Induction) or Sub-Study 2 (Pivotal Induction).
* 12-week Sub-Study 3 (Extended Induction for non-responders).
* 6 weeks (45 days) follow-up period for participants who do not enroll into the Pivotal Maintenance Study (EFC18327). The treatment duration will be up to 12 weeks in each sub-study.

The number of scheduled study visits for participants who continue to the Pivotal Maintenance Study (EFC18327) will be up to 8 (Sub-Study 1 and Sub-Study 2) and up to 15 for participants who enroll in Sub-Study 3.

ELIGIBILITY:
Inclusion Criteria:

Participants aged ≥18 and ≤80 years of age at Screening. Where permitted locally, participants 16 to <18 years of age who meet the definition of Tanner Stage 5 for development

Confirmed diagnosis of moderately to severely active Crohn's Disease (CD) for at least 3 months prior to baseline

Demonstrated inadequate response, have shown loss of response or intolerance to conventional therapies or advanced therapies (ATs)

Exclusion Criteria:

Participants with Ulcerative Colitis (UC) or indeterminate colitis

Participants with two entire missing segments of the: terminal ileum, right colon transverse colon, sigmoid and left colon, and rectum

Prior or current high-grade gastrointestinal (GI) dysplasia

Participants on treatment with but not on stable doses of conventional therapy prior to baseline

Participants receiving prohibited medications or therapies

Participants with previous exposure to anti-TL1A investigational therapy

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-05-14 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
Sub-Study 2: Co-primary endpoints US/FDA: Proportion of participants achieving clinical remission per Crohn's Disease Activity Index (CDAI) at Week 12 | Week 12
  Clinical Remission by CDAI: CDAI score <150. The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease.
Sub-Study 2: Co-primary endpoints US/FDA: Proportion of participants achieving endoscopic response (Simple Endoscopic Score for Crohn's Disease [SES-CD]) at Week 12 | Week 12
  Endoscopic Response is defined as decrease in SES-CD ≥50% from baseline (or a decrease of at least 2 points for participants with a baseline score of 4 or more, and isolated ileal disease) based on central reading. The SES-CD is a standardized method for evaluating disease activity. The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores represent more severe disease.
Sub-Study 2: Co-primary endpoints EU/EMA: Proportion of participants achieving clinical remission per 2-item patient-reported outcome (PRO-2) at Week 12 | Week 12
  Clinical Remission per PRO-2: average daily stool frequency (SF) ≤3 and not worse than the Baseline, and average daily abdominal pain (AP) ≤1 and not worse than the Baseline.
Sub-Study 2: Co-primary endpoints EU/EMA: Proportion of participants achieving endoscopic response (SES-CD) at Week 12 | Week 12
  Endoscopic Response is defined as decrease in SES-CD ≥50% from baseline (or a decrease of at least 2 points for participants with a baseline score of 4 or more, and isolated ileal disease) based on central reading. The SES-CD is a standardized method for evaluating disease activity. The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores represent more severe disease.

SECONDARY OUTCOMES:
Sub-Study 2: Proportion of participants achieving CDAI clinical response at Week 12 | Week 12
  CDAI clinical response is defined as decrease in CDAI score of 100 points or more from baseline.
Sub-study 2: Proportion of participants achieving CDAI clinical response and endoscopic response (SES-CD) at Week 12 | Week 12
  CDAI clinical response is defined as decrease in CDAI score of 100 points or more from baseline. Endoscopic Response by SES-CD was defined as a decrease in SES-CD ≥50% from baseline (or a decrease of at least 2 points for participants with a baseline score of 4 or more, and isolated ileal disease) based on central reading.
Sub-study 2: Proportion of participants achieving endoscopic SES-CD remission at Week 12 | Week 12
  Endoscopic Remission by SES-CD is defined as SES-DC ≤4 points (SES-CD ≤2 points for isolated ileal disease) and a SES-CD decrease ≥2 points with no SES-CD sub score >1 point from baseline
Sub-study 2: US/FDA: Proportion of participants achieving clinical remission per PRO-2 at Week 12 | Week 12
  Clinical Remission per PRO-2: average daily SF ≤3 and not worse than the Baseline, and average daily AP ≤1 and not worse than the Baseline.
Sub-study 2: EU/EMA: Proportion of participants achievingclinical remission per CDAI at Week 12 | Week 12
  Clinical Remission by CDAI: CDAI score <150. The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease.
Sub-study 2: Proportion of participants achieving ulcer-free endoscopy (in the subset of participants with ulcers at baseline) at Week 12 | Week 12
  Ulcer-free endoscopy: SES-CD ulcerated surface sub-score of 0 in participants with SES-CD ulcerated surface sub-score ≥1 at Baseline, as scored by a central reader.
Sub-study 2: Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue Short Form 7a T-score at Week 12 | Baseline, Week 12
  The PROMIS Fatigue Short Form 7a uses a 5-point Likert scale for each of its 7 items, resulting in a raw score range of 7 to 35. This raw score is then converted into a T-score, with a mean of 50 and a standard deviation of 10, based on US national norms. Higher T-scores indicate greater fatigue.
Sub-study 2: Proportion of participants achieving CDAI clinicalresponse at Week 4 | Week 4
  CDAI clinical response is defined as decrease in CDAI score of 100 points or more from baseline.
Sub-study 2: US/FDA: Proportion of participants achievingcorticosteroid free remission (in the subset ofparticipants with corticosteroids at baseline) perCDAI at Week 12 | Week 12
  Corticosteroid free remission per CDAI: proportion of participants who discontinue corticosteroid use for CD and achieve clinical remission per CDAI (CDAI score <150) at Week 12, in participants taking corticosteroids for CD at Baseline.
Sub-study 2: EU/EMA: Proportion of participants achievingcorticosteroid free remission per PRO-2 (in thesubset of participants with corticosteroids atbaseline) at Week 12 | Week 12
  Corticosteroid free remission by PRO-2: proportion of participants who discontinue corticosteroid use for CD and achieve clinical remission per PRO-2 (average daily SF ≤3 and not worse than the baseline, and average daily AP ≤1 and not worse than the baseline) at Week 12, in participants taking corticosteroids for CD at Baseline.
Sub-study 2: Proportion of participants achieving CDAI clinical remission and endoscopic remission (SES-CD) at Week 12 | Week 12
  Clinical Remission by CDAI: CDAI score <150. Endoscopic Remission: SES-CD ≤4 points (SES-CD ≤2 points for isolated ileal disease) and a SES-CD decrease ≥2 points with no SES-CD sub score >1 point from baseline.
Sub-study 2: Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) total score at Week 12 | Baseline, Week 12
  IBDQ instrument consist of 32 items exploring 4 dimensions: "bowel symptoms" (10 items), "systemic symptoms" (5 items), "emotional function" (12 items) and "social function" (5 items). The total IBDQ total score ranges from 32 to 224 with higher score indicating better quality of life.
Sub-study 2: Proportion of participants with no bowel urgency byNumeric Rating Scale (NRS) at Week 12 | Week 12
  The NRS for bowel urgency is a well-defined and reliable instrument to evaluate treatment benefits in participants with CD. The NRS for bowel urgency measures the severity of bowel urgency-the sudden or immediate need to have a bowel movement-experienced in the past 24 hours. This tool utilizes an 11-point scale for evaluation, from 0 (no urgency) to 10 (worst possible urgency).
Sub-study 2: Proportion of participants with CD-related hospitalizations by Week 12 | Baseline through Week 12
Sub-study 2: Number of participants with any Treatment Emergent Adverse Events (TEAEs), TEAE of special interest (TEAESIs), TE serious adverse event (TESAEs), and TEAEs leading to permanent study intervention discontinuation | Baseline through 45 days after the last dose
Sub-study 2: Serum concentrations of duvakitug | Baseline to Week 12
Sub-study 2: Incidence of treatment-emergent Anti-drug Antibodies (ADA) against duvakitug | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (71):
- United States (60):
  - Onyx Clinical Research - Site Number: 8400021, Peoria, Arizona
  - Del Sol Research Management, LLC: 8400012, Tucson, Arizona
  - Preferred Research Partners: 8400018, Little Rock, Arkansas
  - Kagoshima IBD Gastroenterology Clinic - Site Number: 8400008, Canoga Park, California
  - Southern California GI & Liver Centers: 8400062, Coronado, California
  - GMC Clinical Research, LLC: 8400113, Folsom, California
  - TLC Clinical Research Inc.: 8400030, Los Angeles, California
  - United Medical Doctors CA: 8400044, Murrieta, California
  - Prospective Research Innovations Inc.: 8400017, Rancho Cucamonga, California
  - Valiance Clinical Research - Tarzana: 8400023, Tarzana, California
  - Clinical Trials Management Services: 8400047, Thousand Oaks, California
  - Amicis Research Center-Valencia: 8400064, Valencia, California
  - Om Research, LLC - Victorville - Site Number: 8400022, Victorville, California
  - Peak Gastroenterology Associates - Colorado Springs: 8400039, Colorado Springs, Colorado
  - Precision Clinical Research: 8400059, Coral Springs, Florida
  - Sarkis Clinical Trials-Ocala: 8400048, Gainesville, Florida
  - Clinical Research of Osceola: 8400013, Kissimmee, Florida
  - Columbus Clinical Services LLc: 8400038, Miami, Florida
  - Regis Clinical Research, LLC-Site Number: 8400041, Miami, Florida
  - Bio Research Partner: 8400053, Miami, Florida
  - Correa Research Center-Site Number: 8400010, Miami, Florida
  - NMC Research LLC - Site Number: 8400033, Tampa, Florida
  - M3 Wake Research - Atlanta: 8400028, Sandy Springs, Georgia
  - EBGS Clinical Research Center, LLC: 8400037, Snellville, Georgia
  - GI Alliance - Glenview - Site Number: 8400068, Glenview, Illinois
  - Illinois Gastroenterology Group d/b/a GI Alliance - Gurnee - Site Number: 8400049, Gurnee, Illinois
  - Gastroenterology Health Partners, PLLC - Site Number: 8400100, New Albany, Indiana
  - GI Alliance - Baton Rouge - Site Number: 8400129, Baton Rouge, Louisiana
  - GI Alliance - Metairie: 8400124, Metairie, Louisiana
  - Delta Research Partners: 8400087, Monroe, Louisiana
  - Mid-Atlantic GI Research, LLC - Site Number: 8400106, Greenbelt, Maryland
  - Gastroenterology Associates of Western Michigan - Site Number: 8400060, Wyoming, Michigan
  - Gateway Gastroenterology: 8400097, Chesterfield, Missouri
  - BVL Clinical Research: 8400005, Liberty, Missouri
  - Premier Health Research, LLC - Site Number: 8400114, Sparta, New Jersey
  - MedTraits NY: 8400045, Maspeth, New York
  - Manhattan Clinical Research, LLC - Site Number: 8400069, New York, New York
  - New York Gastroenterology Associates: 8400009, New York, New York
  - OnSite Clinical Solutions: 8400051, Charlotte, North Carolina
  - Cross Creek Medical Clinic: 8400057, Fayetteville, North Carolina
  - Monroe Biomedical Research - Site Number: 8400046, Monroe, North Carolina
  - ClinTrial Research, LLC - Site Number: 8400043, Raleigh, North Carolina
  - Plains Medical Clinic: 8400078, Fargo, North Dakota
  - Ohio Gastroenterology Group Inc.: 8400006, Columbus, Ohio
  - DSI Research, LLC: 8400115, Dayton, Ohio
  - DSI Research, LLC - Site Number: 8400105, Springboro, Ohio
  - North Shore Gastroenterology Research - Site Number: 8400130, Westlake, Ohio
  - Central Sooner Research: 8400094, Norman, Oklahoma
  - University Gastroenterology - GI Alliance - Site Number: 8400103, Providence, Rhode Island
  - Biocentric Health Research Partner: 8400089, West Columbia, South Carolina
  - Tri-Cities Gastroenterology: 8400076, Kingsport, Tennessee
  - Valley Institute of Research: 8400004, Harlingen, Texas
  - Innovare Research Group: 8400067, Lake Jackson, Texas
  - Texas Digestive Disease Consultants dba GI Alliance - Lubbock - Site Number: 8400092, Lubbock, Texas
  - Texas Digestive Disease Consultants, PLLC. dba GI Alliance - Southlake - Site Number: 8400101, Southlake, Texas
  - Texas Gastro Consultants: 8400029, Tomball, Texas
  - Tyler Research Institute, LLC: 8400095, Tyler, Texas
  - Blue Ridge Medical Research: 8400020, Lynchburg, Virginia
  - Clinical Research Partners - Site Number: 8400080, Richmond, Virginia
  - The Vancouver Clinic Inc. P.S. - Site Number: 8400090, Vancouver, Washington
- Canada (3):
  - Investigational Site Number: 1240009, Hamilton
  - Investigational Site Number: 1240010, Oakville
  - Investigational Site Number: 1240003, Toronto
- Japan (7):
  - Kagoshima IBD Gastroenterology Clinic Site Number : 3920049, Kagoshima
  - Ofuna Chuo Hospital: 3920029, Kamakura
  - Kokikai Tsujinaka Hospital Kashiwanoha: 3920031, Kashiwa
  - Aoyama Clinic: 3920018, Kobe
  - Sapporo Tokushukai Hospital: 3920019, Sapporo
  - Tokai University Hachioji Hospital: 3920030, Tokyo
  - Toyama University Hospital: 3920032, Toyama
- Wellness Clinical Research - Vega Baja: 8400099, Vega Baja, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC18326 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26861&tenant=MT_SNY_9011